CLINICAL TRIAL: NCT02349464
Title: Promoting Lactation Education, Access, and Support Efforts for Preterm Infants
Acronym: PLEASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR#27878
Record Dates: First submitted 2015-01-15; First posted 2015-01-29 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): For infants receiving pediatric care at one of the seven intervention practices, mothers will receive the Specialized Preterm Infant/Mother Dyad Lactation Support which includes home equipment and pediatric clinic-lactation support to support lactation for four months post-hospital discharge.
  Interventions: Other: Specialized Preterm Infant/Mother Dyad Lactation Support
- Control (No Intervention): For infants receiving pediatric care at one of the seven control practices, mothers will receive standard support.

INTERVENTIONS:
Other: Specialized Preterm Infant/Mother Dyad Lactation Support — Mother will receive home equipment and pediatric clinic lactation support.
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine whether a post-hospital discharge lactation support system increases preterm infant intake of mother's milk.

DETAILED DESCRIPTION:
Preterm infants have barriers to successful breastfeeding that include oral feeding immaturity and high nutritional needs. Therefore, successful preterm infant breastfeeding requires increased counseling and equipment support compared to full-term infant breastfeeding. Inpatient preterm infant care has responded to these barriers, with specialized preterm infant lactation support. Unfortunately, for preterm infants, the onset of feeding maturity often coincides with hospital discharge and, therefore, inpatient, specialized lactation support ends just as the infant initiates nutritive feeding at the breast. Therefore, the success of preterm infant breastfeeding relies on the home environment and the community pediatric caregivers. A program has been created to provide this specialized preterm infant/mother outpatient lactation support. The program includes in-home availability of a hospital-grade electric pump and an infant weigh scale and pediatric clinic-based lactation counseling support. Fourteen pediatric practices are included in this study. Seven practices were randomized to intervention and seven were randomized to be controls.

ELIGIBILITY:
Inclusion Criteria:

* Any infant discharge to home from the Medical University of South Carolina neonatal services
* Born <35 weeks' gestation
* Mother providing her milk and plans to continue providing her milk for at least 6 months
* The infant's post-discharge pediatric clinic identified by mother as one involved in the study
* The eligible twin will be the first twin discharged from the hospital or, if discharge occurs simultaneously, the infant identified in the hospital as "twin A" will be eligible.

Exclusion Criteria:

* Infants with major congenital anomalies
* Infants with anomalies affecting oral intake
* Infants receiving tube feeds at hospital discharge
* Infants receiving parenteral nutrition at hospital discharge
* Triplet or greater pregnancies
* Twin of the one enrolled twin will not be eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-12; Primary Completion 2018-02 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Preterm infant intake of mother's milk post-hospital discharge measured by survey. | 4 months

SECONDARY OUTCOMES:
Preterm infant breastfeeding post-hospital discharge measured by survey. | 4 months
Sustaining preterm infant mother's milk intake post-hospital discharge measured by survey. | 6 months
Preterm infant growth post-hospital discharge collected from pediatric clinic medical record. | 6 months
Preterm infant re-hospitalization post-hospital discharge collected from pediatric clinic medical record. | 6 months
Preterm infant respiratory illness events post-hospital discharge collected from pediatric clinic medical record. | 6 months
Preterm infant gastrointestinal illness events post-hospital discharge collected from pediatric clinic medical record. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sarah N Taylor, MD, MSCR, Principal Investigator — Medical University of South Carolina